CLINICAL TRIAL: NCT04533802
Title: Personality and Genotypic Markers That Predict Individual Differences in Susceptibility to Stress-induced Alcohol Misuse: a Feasibility Study.
Brief Title: Risk Factors for Stress-induced Alcohol Misuse: Genetic Predictors and Mediation by Personality Type
Acronym: RISK
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/63
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-01

CONDITIONS: Alcohol Use, Unspecified
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To examine whether variation in 'risk-taking' personality and linked genetic variants predicts susceptibility to, and resilience against, stress-induced alcohol misuse.

DETAILED DESCRIPTION:
Alcohol misuse is a global health issue responsible for over 1 million hospital admissions per annum in the UK with a combined cost of approximately £21 billion. Chronic alcohol misuse in patients who attend hospital for alcohol-related illness/injury is common, with relapse and recidivism almost ubiquitous. Patients often report that 'stress' was a catalyst for their drinking episodes, but we do not know exactly who is most at risk, how stress leads to drinking, or the genetic basis for this risk. This research aims to seek to identify patients at higher risk of stress-induced alcohol misuse, or who are more resilient to stress in this context, using a combination of analyses ranging from genetic variants to personality tests and clinical follow-up. The ultimate goal is that patients engaging with alcohol services can receive personalised and focussed treatment and enhance recovery

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged (min) 18 years
* Attended Portsmouth Hospitals University Trust following illness/injury related to alcohol use
* Has a maximum AUDIT score of 15
* Is willing and able to comply with study procedures
* Willing and able to give informed consent for participation in the study.
* Must be recruited within 24 hrs of ASNS referral, and able to be tested within 48 hours of referral

Exclusion Criteria:

ny reported/suspected intellectual/learning disabilities (e.g., Down's Syndrome), neurodevelopmental disorders (e.g., Autism, Asperger's) or acquired brain injury

* Has previously participated in this study
* Should not be under the influence of alcohol during the study (12hrs previous to taking part) - to be determined via breathalyser.
* Any history of advanced liver disease (clinical diagnosis of cirrhosis, jaundice, encephalopathy, ascites, variceal haemorrhage)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be patients attending Portsmouth Hospitals University Trust following alcohol-related illness/injury and an AUDIT score of greater than 15 (suggesting high risk of dependence and alcohol misuse). They will be adults (>18 years).
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Alcohol misuse | immediately after the procedure
  Measured using the alcohol use disorders identification test (AUDIT) (higher the score the worse the outcome)
Recent stressors | Immediately after the study visit
  Measured using the 30 item Stress Overload Scale questionnaire (higher the score, the worse the outcome)
Life Events | Immediately after the study visit
  Measured using the Life Events Checklist Questionnaire (the higher the score the worse the outcome)
Impulse Behaviour | Immediately after the study visit
  Measured using the the Urgency, Premeditation (lack of), Perseverance (lack of), Sensation Seeking, Positive Urgency, Impulsive Behavior Scale (UPPS-P) higher values indicate more impulsive behavior.
Risk taking behaviour | Immediately after the study visit
  Measured by the Stop Signal Reaction Time Task (computer task) which measures the ability to inhibit a planned response
Molecular Anaylsis | Immediately after the study visit
  Cheek swabs will be taken from all participant to carry out genomic DNA analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth University Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No